CLINICAL TRIAL: NCT03583242
Title: Multimodal Image Study of Retinal Inflammation Markers After Corticoid and Antiangiogenic Treatment in Pacients With Diabetic Macular Edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Other Study IDs: IIBSP-RET-2018-13
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Angiogenesis Inhibitors; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DME treat with antiangiogenic: * 3 Intravitreal injections of 0.05 ml of Aflibercept (40 mg/ml) during 3 months (one per month) The clinical management of the patients will be adapted to the treatment standards of the Ophthalmology Service of the Hospital de la Santa Creu and Sant Pau, without the realization of this study influencing such process.
  * 1 Injection of dexamethasone intravitreal implant 0.7mg. The clinical management of the patients will be adapted to the treatment standards of the Ophthalmology Service of the Hospital de la Santa Creu and Sant Pau, without the realization of this study influencing such process.
  Interventions: Drug: Antiangiogenic Agents; Drug: Corticosteroid

INTERVENTIONS:
Drug: Antiangiogenic Agents — 3 Intravitreal injections of 0.05 ml of Aflibercept (40 mg/ml) during 3 months (one per month) The clinical management of the patients will be adapted to the treatment standards of the Ophthalmology Service of the Hospital de la Santa Creu and Sant Pau, without the realization of this study influencing such process.
Drug: Corticosteroid — 1 Injection of dexamethasone intravitreal implant 0.7mg. The clinical management of the patients will be adapted to the treatment standards of the Ophthalmology Service of the Hospital de la Santa Creu and Sant Pau, without the realization of this study influencing such process.

SUMMARY:
* Main objective: Inflammation factors in imaging techniques of diabetic macular edema
* Prospective observational design
* Disease under study: Diabetic macular edema
* Methodology: Collection of the image data in the usual control (baseline visit, 4th month)
* Population under study and total number of subjects Diabetics with macular edema.
* Approximate N: 80 pacients.
* Expected duration of the study: 12 months.

DETAILED DESCRIPTION:
PROBLEM STATEMENT:

Background Currently the DME (diabetic macular edema) can be treated with 2 types of intravitreous treatment: corticosteroids (Ozurdex) or antiangiogenic (Eylea). Until a few years ago it was treated with photocoagulation. But the most rapid advances have been made at the level of image tests with more and more cutting-edge OCTs (optical coherence tomography) that allow an image of better quality and precision allowing more and more details to be observed. Also the new photographs of autofluorescences or the Angio-OCT allow to observe many more details. Therefore this recent field in constant progression remains unexplored. Current studies on inflammation factors before and after treatment are few and with small N that do not exceed 20.

This study aims to observe all these inflammation factors of images, anatomical involvement by DME and see how they respond after intravitreal treatment. As another more pretentious objective would be to draw some conclusion about the drugs used according to the changes observed in the images.

Justification Today, these multiple imaging techniques are the only way to obtain information about DME apart from the direct exploration of the fundus, the changes they produce and the responses to treatment. Since its appearance, the management and follow-up of patients affected by DME has been constantly improved. Given the constant evolution of the quality of the images the investigators must study the new possibilities that they offer us.

Investigation questions What are the changes in inflammatory markers that can be detected by multimodal study of new imaging techniques before and after corticosteroid and antiangiogenic treatment in patients with diabetic macular edema?

OBJECTIVE OF THE STUDY:

To study changes in inflammation markers by multimodal study of new imaging techniques after corticosteroid and antiangiogenic treatment in patients with diabetic macular edema

- Definition of variables

Main variable:

- Markers of image inflammation: choroidal thickness, central macular thickness, type of DME, disruption of the ellipsoid line, disruption of the external limiting membrane, disorganization of retinal inner layers, number of hyperreflective points, presence of hyperautofluorescent lesions, presence of epiretinal membrane.

These markers will be evaluated before treatment and 4 months after treatment to observe the changes that have occurred.

Other variables to be collected:

* Demographic data: sex, age
* Pathological antecedents: Degree of diabetic retinopathy, type of DM, last HbA1c, DM evolution time.
* HbA1c: last value that the patient has in his usual follow-up.

Size of the expected sample Approx N = 80 A formal calculation of the sample size has not been made. It is considered that with an N of 80 it will be sufficient to achieve the objectives of the study.

METHODOLOGY: Information sources Patients will be recruited from the Ophthalmology service in the different Retina offices of the Hospital de la Santa Creu i Sant Pau.

In case of fulfilling the selection criteria and accepting to participate by signing the informed consent, the necessary information will be collected from the clinical history.

The usual tests (visual acuity, OCT, angio-OCT, retinographies, autofluorescence) will be carried out and the usual treatment will be indicated (intravitreal injections of Eylea or Ozurdex) After 4 months of treatment at the usual monitoring visit, the same usual tests will be performed (visual acuity, OCT, angio-OCT, retinographies, autofluorescence). After that, the study with the patient ends.

As indicated, the treatment and screening methods are those that are routinely performed in the center to patients with this pathology, so it does not imply additional requests or potential risks from the present study.

- Management and Analysis of data: Management and analysis of the data with the SPSS statistical program and with the help of the Hospital's Biostatistics service.

QA The researcher will guarantee the accuracy and integrity of the data, as well as all the reports that are required.

The researcher will save the study documents until at least 5 years after completion of the study.

Upon the request of the monitor, auditor, CEIC or health authority, the researcher will have available all the files related to the study, allowing direct access to the data or source documents for the realization of the monitoring, the audit, the review by the CEIC , as well as the inspection of the trial by the competent authorities.

ETHICAL ASPECTS:

Benefit-risk evaluation of the research No risks arising from participation are expected, since the usual practice of treatment is not changed and no image test is toxic or has side effects.

Ethical considerations, about information to subjects and informed consent The study will be carried out strictly following the international ethical recommendations for medical research in humans. The researcher will be responsible for ensuring that the study is conducted in accordance with the standards set out in the Declaration of Helsinki.

Before starting the study, the Ethical Committee of the Hospital of Santa Creu i Sant Pau (CEIC) must approve the protocol of the study, the information that will be given to the subject and the model of informed consent that will be used.

The CEIC will be informed of any amendment subsequent to the protocol and its opinion should be requested in case a new evaluation of the ethical aspects of the study is necessary.

It is the researcher's responsibility to obtain the informed consent of the patient. The patient will not be able to participate in any specific procedure of the study before obtaining their consent, or that of their legal / family tutor when the patient is not able to give their consent for their clinical situation.

Before including any subject in the study and before obtaining the informed consent, the researcher or the person designated by the same, will explain to the possible participant subject or their legal / family tutor, the objectives, methods and potential risks of the study and any annoyance that this may cause. The explanation about the nature, scope and possible consequences of the study will be made in an understandable language.

The potential participant or his / her legal / family tutor must have time to reflect on their decision to participate in the study, and have the opportunity to ask questions. After this explanation, and before entering the study, the consent must be properly recorded by the signature of the subject or legal / family tutor.

Confidentiality of the data:

Regarding the confidentiality of the study data, the provisions of Organic Law 15/1999 of December 13, on "Protection of Personal Data" will be followed.

Interference with the doctor's prescription habits:

The clinical management of the patients will be adapted to the treatment standards of the Ophthalmology Service of the Hospital de la Santa Creu and Sant Pau, without the realization of this study influencing such process.

PLANS FOR THE DISSEMINATION OF RESULTS:

Dissemination of the results in publications of medical journals and for the realization of the doctoral thesis

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of diabetic macular edema
* Without any intravitreal treatment during the last three months
* Patients who require intravitreal corticoid or antiangiogenic treatment following the usual clinical practice

Exclusion Criteria:

* Any other macular pathology ( for exemple age-related macular degeneration)
* Proliferative diabetic retinopathy
* Any other eye involvement that may influence visual acuity (eg, uncontrolled glaucoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient adult with diabetic macular edema in external consultations of our department that require intravitravitreal treatment according to daily clinical practice and that satisfy inclusion an exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Macular thickness | At first visit and 4 months after the first intravitreal injection
  Measured by OCT in micrometer
Coroidal thickness | At first visit and 4 months after the first intravitreal injection
  Measured by OCT (EDI mode) in micrometer
Numbers of hyperreflective intraretinal spots | At first visit and 4 months after the first intravitreal injection
  Measured by OCT scans
Increased macular autofluorescence | At first visit and 4 months after the first intravitreal injection
  Autofluorescence of the fundus

SECONDARY OUTCOMES:
Best corrected visual acuity | At first visit and 4 months after the first intravitreal injection
  Visual acuity test: ETDRS at 4 meters
Type of diabetic macular edema | At first visit and 4 months after the first intravitreal injection
  Direct visualization with OCT images: cystic, subretinal fluid, spongiform
Presence of epiretinal membrane | At first visit and 4 months after the first intravitreal injection
  Direct visualization with OCT images
Disruption of ellipsoid line and external limiting membrane | At first visit and 4 months after the first intravitreal injection
  Direct visualization with OCT images
Disorganization of the retinal inner layers | At first visit and 4 months after the first intravitreal injection
  Direct visualization with OCT images
Subfoveal neuroretinal detachment | At first visit and 4 months after the first intravitreal injection
  Direct visualization with OCT images

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vujosevic S, Torresin T, Berton M, Bini S, Convento E, Midena E. Diabetic Macular Edema With and Without Subfoveal Neuroretinal Detachment: Two Different Morphologic and Functional Entities. Am J Ophthalmol. 2017 Sep;181:149-155. doi: 10.1016/j.ajo.2017.06.026. Epub 2017 Jul 4. PMID 28687219
- [Background] Murakami T, Suzuma K, Dodo Y, Yoshitake T, Yasukura S, Nakanishi H, Fujimoto M, Oishi M, Tsujikawa A. Decorrelation Signal of Diabetic Hyperreflective Foci on Optical Coherence Tomography Angiography. Sci Rep. 2018 Jun 11;8(1):8798. doi: 10.1038/s41598-018-27192-9. PMID 29892079
- [Background] Santos AR, Costa MA, Schwartz C, Alves D, Figueira J, Silva R, Cunha-Vaz JG. OPTICAL COHERENCE TOMOGRAPHY BASELINE PREDICTORS FOR INITIAL BEST-CORRECTED VISUAL ACUITY RESPONSE TO INTRAVITREAL ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR TREATMENT IN EYES WITH DIABETIC MACULAR EDEMA: The CHARTRES Study. Retina. 2018 Jun;38(6):1110-1119. doi: 10.1097/IAE.0000000000001687. PMID 28613220
- [Background] Kim TK, Shin HY, Kim SY, Lee YC, Lee MY. Factors Influencing Intravitreal Bevacizumab and Triamcinolone Treatment in Patients with Diabetic Macular Edema. Eur J Ophthalmol. 2017 Nov 8;27(6):746-750. doi: 10.5301/ejo.5000974. PMID 28430331
- [Background] Fickweiler W, Schauwvlieghe AME, Schlingemann RO, Maria Hooymans JM, Los LI, Verbraak FD; BRDME Research Group. PREDICTIVE VALUE OF OPTICAL COHERENCE TOMOGRAPHIC FEATURES IN THE BEVACIZUMAB AND RANIBIZUMAB IN PATIENTS WITH DIABETIC MACULAR EDEMA (BRDME) STUDY. Retina. 2018 Apr;38(4):812-819. doi: 10.1097/IAE.0000000000001626. PMID 28406860
- [Background] Chakravarthy U, Yang Y, Lotery A, Ghanchi F, Bailey C, Holz FG, Downey L, Weber M, Eter N, Dugel PU. CLINICAL EVIDENCE OF THE MULTIFACTORIAL NATURE OF DIABETIC MACULAR EDEMA. Retina. 2018 Feb;38(2):343-351. doi: 10.1097/IAE.0000000000001555. PMID 28257378
- [Background] Seo KH, Yu SY, Kim M, Kwak HW. VISUAL AND MORPHOLOGIC OUTCOMES OF INTRAVITREAL RANIBIZUMAB FOR DIABETIC MACULAR EDEMA BASED ON OPTICAL COHERENCE TOMOGRAPHY PATTERNS. Retina. 2016 Mar;36(3):588-95. doi: 10.1097/IAE.0000000000000770. PMID 26398695